CLINICAL TRIAL: NCT04197934
Title: Phase I Study to Evaluate Safety, Tolerability, Pharmacokinetics and Anti-Tumor Activity of WSD0922-FU
Brief Title: WSD0922-FU for the Treatment of Glioblastoma, Anaplastic Astrocytoma, or Non-small Cell Lung Cancer With Central Nervous System Metastases
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1914; R01FD007288 (FDA); NCI-2019-07825 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1914 (Other: Mayo Clinic); 19-005001 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2019-11-25; First posted 2019-12-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Anaplastic Astrocytoma, IDH-Wildtype; Glioblastoma, IDH-Wildtype; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Malignant Neoplasm in the Central Nervous System; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose escalation (WSD0922-FU) (Experimental): Patients receive WSD0922-FU PO QD or BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, MRI, and blood sample collection on study. Patients with NSCLC with LM also undergo collection of CSF samples on study.
  Interventions: Procedure: Biospecimen Collection - blood samples; Procedure: Biospecimen Collection - CSF samples; Procedure: Computed Tomography; Drug: EGFR/EGFRvIII Inhibitor WSD0922-FU; Procedure: Magnetic Resonance Imaging
- Dose expansion Cohort I (WSD0922-FU) (Experimental): Patients with GBM/AA receive WSD0922-FU PO on days 1 and 4 of cycle 0. Patients then receive WSD0922-FU PO BID on days 1-28 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI during screening and on study, as well as blood sample collection on study. Patients may undergo additional optional blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection - blood samples; Drug: EGFR/EGFRvIII Inhibitor WSD0922-FU; Procedure: Magnetic Resonance Imaging
- Dose expansion Cohort II (WSD0922-FU, surgery) (Experimental): Patients with BTP receive a single dose of WSD0922-FU prior to surgery. Patients then undergo surgical resection of brain tumor. After surgery, patients receive WSD0922-FU PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI during screening and on study, as well as blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection - blood samples; Drug: EGFR/EGFRvIII Inhibitor WSD0922-FU; Procedure: Magnetic Resonance Imaging; Procedure: Therapeutic Conventional Surgery
- Dose expansion Cohort III (WSD0922-FU) (Experimental): Patients with NSCLC receive WSD0922-FU PO BID on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI and CT during screening and on study, as well as blood sample collection on study. Patients with LM also undergo collection of CSF samples on study. Patients may also undergo optional blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection - blood samples; Procedure: Biospecimen Collection - CSF samples; Procedure: Computed Tomography; Drug: EGFR/EGFRvIII Inhibitor WSD0922-FU; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection - blood samples — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Biospecimen Collection; Specimen Collection
Procedure: Biospecimen Collection - CSF samples — Undergo collection of CSF samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Biospecimen Collection; Specimen Collection
  Arms: Dose escalation (WSD0922-FU); Dose expansion Cohort III (WSD0922-FU)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
  Arms: Dose escalation (WSD0922-FU); Dose expansion Cohort III (WSD0922-FU)
Drug: EGFR/EGFRvIII Inhibitor WSD0922-FU — Given PO
  Other Names: BBB Penetrable EGFR/EGFRvIII Inhibitor WSD0922-FU; EGFR Mutant Inhibitor WSD0922-FU; WSD 0922-FU; WSD-0922-FU; WSD0922-FU
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Therapeutic Conventional Surgery — Undergo surgical resection
  Arms: Dose expansion Cohort II (WSD0922-FU, surgery)

SUMMARY:
This phase I trial studies the side effects and best dose of WSD0922-FU for the treatment of glioblastoma, anaplastic astrocytoma, or non-small cell lung cancer that has spread to the central nervous system (central nervous system metastases). WSD0922-FU is a targeted treatment which blocks the EGFR protein - a strategy that has led to a lot of benefit in patients with many different cancers. WSD0922-FU may also be able to get into cancers in the brain and spinal cord and help patients with brain and spinal cord cancers.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose (MTD) and/or the recommended phase 2 dose (RP2D) of EGFR/EGFRvIII inhibitor WSD0922-FU (WSD0922-FU) in subjects with recurrent glioblastoma, IDH wildtype (GBM), anaplastic astrocytoma, IDH wildtype (AA) and central nervous system (CNS) metastases of non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To evaluate the incidence of treatment-emergent adverse events (TEAEs) related to WSD0922-FU.

II. To assess anti-tumor activity: intracranial and extracranial overall response rate (ORR), and change in tumor size compared with baseline according to Response Assessment in Neuro-Oncology (RANO) criteria for GBM/AA and Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for NSCLC.

III. To assess anti-tumor activity: intracranial and extracranial disease control rate (DCR) and change in tumor size compared with baseline according to RANO criteria for GBM/AA and RECIST 1.1 for NSCLC.

IV. To assess anti-tumor activity: intracranial and extracranial duration of response (DOR) and change in tumor size compared with baseline according to RANO criteria for GBM/AA and RECIST 1.1 for NSCLC.

V. To assess anti-tumor activity: intracranial and extracranial progression-free survival (PFS) and change in tumor size compared with baseline according to RANO criteria for GBM/AA and RECIST 1.1 for NSCLC.

EXPLORATORY/CORRELATIVE RESEARCH OBJECTIVES:

I. To investigate the presence and/or identity of the drug metabolites of WSD0922-FU, and the concentrations of these in the plasma, cerebrospinal fluid (CSF), and tumor.

II. To assess plasma concentration of WSD0922-FU and metabolite SN16110801P1 and pharmacokinetics (PK) parameters after single and multiple doses of WSD0922-FU.

III. To assess the brain tumor pharmacokinetics of WSD0922-FU and SN16110801P1 after a single dose of WSD0922-FU (Dose Expansion - Brain tumor penetration [BTP] cohort only).

IV. To assess cerebrospinal fluid (CSF) concentration of WSD0922-FU and SN16110801P1 after multiple doses of WSD0922-FU (Dose Expansion - NSCLC cohort only).

V. To explore the impact of tumor markers (e.g. MGMT promoter methylation, EGFR mutation [including EGFR vIII], PTEN deletion, TP53 mutation, etc.) on clinical parameters associated with WSD0922-FU treatment.

VI. To evaluate and measure pharmacodynamic biomarkers of inhibition of EGFR and downstream signals in tumor samples after a single dose of WSD0922-FU (Dose Expansion Cohort - BTP cohort only).

VII. To evaluate the effect of food on the pharmacokinetics of single dose of WSD0922-FU in plasma (Dose Expansion - GBM/AA cohort only).

OUTLINE: This is a dose-escalation study.

DOSE ESCALATION: Patients receive WSD0922-FU orally (PO) once daily (QD) or twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT), magnetic resonance imaging (MRI), and collection of blood samples on study. Patients with NSCLC with leptomeningeal metastases (LM) also undergo collection of CSF samples on study.

DOSE EXPANSION: Patients are assigned to 1 of 3 cohorts.

COHORT I: Patients with GBM/AA receive WSD0922-FU PO on days 1 and 4 of cycle 0. Patients then receive WSD0922-FU PO BID on days 1-28 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI during screening and on study, as well as blood sample collection on study. Patients may undergo additional optional blood sample collection on study.

COHORT II: Patients with BTP receive a single dose of WSD0922-FU prior to surgery. Patients then undergo surgical resection of brain tumor. After surgery, patients receive WSD0922-FU PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI during screening and on study, as well as blood sample collection on study.

COHORT III: Patients with NSCLC receive WSD0922-FU PO BID on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI and CT during screening and on study, as well as blood sample collection on study. Patients with LM also undergo collection of CSF samples on study. Patients may also undergo optional blood sample collection on study.

After completion of study treatment, patients are followed up at 4-6 weeks, then every 2 months until progressive disease, at progressive disease, and then every 3 months after progressive disease for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Pre-Registration - Inclusion Criteria Specific to Dose Escalation Cohort

  * Histolopathological and/or molecular confirmation of either glioblastoma, IDH wildtype (GBM), (as defined by either the 2016 or 2021 World Health Organization [WHO] classifications) anaplastic astrocytoma, IDH wildtype (AA) (as defined by the 2016 WHO classification) or non-small cell lung cancer (NSCLC)
  * EGFR Status:

    * GBM/AA must either EGFR amplification and/or any activating EGFR mutation (e.g. A289T, EGFRvIII , etc.)
    * NSCLC must have a confirmed activating EGFR mutation (e.g. Del19, L858R, EGFRvIII, G719A, L861Q, T790M, C797S, etc.)
* Pre-Registration - Inclusion Criteria Specific to Dose Expansion Cohorts

  * Glioblastoma, IDH wildtype/Anaplastic astrocytoma, IDH wildtype (GBM/AA) Cohort:

    * Diagnosis: Histological or molecular confirmation of either glioblastoma, IDH wildtype (GBM) (as defined by either the 2016 or 2021 WHO classifications) or anaplastic astrocytoma, IDH wildtype (AA) (as defined by the 2016 WHO classification)
    * EGFR status: GBM/AA must have EGFRvIII mutation
  * Brain Tumor Penetration (BTP) Cohort:

    * Diagnosis: Histopathological or molecular confirmation of either glioblastoma, IDH wildtype (GBM) (as defined by either the 2016 or 2021 WHO classifications) or anaplastic astrocytoma, IDH wildtype (AA) (as defined by the 2016 WHO classification)
    * EGFR status: GBM/AA must have been previously demonstrated to have either EGFR amplification and/or any activating EGFR mutation based on any prior resection
  * Non-Small Cell Lung Cancer (NSCLC) cohort:

    * Diagnosis: Histological confirmation of non-small cell lung cancer (NSCLC)
    * EGFR status: NSCLC must have confirmed activating EGFR mutation. Following protocol amendment 7, NSCLC must have EGFR C797S mutation.
* Registration -Inclusion Criteria Specific to Dose Escalation Cohort

  * Previous treatments:

    * Patients with GBM/AA must have been previously treated with radiation and temozolomide
    * Patients with NSCLC must have been previously treated with at least one line of single-agent therapy with an EGFR TKI e.g. gefitinib, erlotinib, afatinib, or osimertinib)
  * Radiographic progression:

    * Patients with GBM/AA must have radiographic progression based on RANO criteria
    * Patients with NSCLC must have new or radiographic progression in the central nervous system (brain metastases and/or leptomeningeal metastases). Positive confirmation of CSF cytology is both necessary and sufficient to define the presence of leptomeningeal metastases for patients in this study. Patients with positive CSF cytology and brain metastases will be categorized as "leptomeningeal metastases."
  * Measurable disease
  * Eastern Cooperative Oncology Group (ECOG) 0 or 1. For patients with NSCLC with leptomeningeal metastases, ECOG 2 is also acceptable
* Registration - Inclusion Criteria Specific to Dose Expansion Cohorts

  * Glioblastoma, IDH wildtype/Anaplastic astrocytoma, IDH wildtype (GBM/AA) Cohort:

    * Previous treatments: Patients must have been previously treated with radiation and temozolomide. First recurrence only (no additional systemic therapies have been administered for recurrent disease)
    * Radiographic progression: Patients with GBM/AA must have radiographic progression based on RANO criteria
    * Patients remain eligible for enrollment if the recurrent disease has been surgically removed
    * Performance status: ECOG 0 or 1
  * Brain Tumor Penetration (BTP) Cohort:

    * Previous treatments: Patients must have been previously treated with radiation and temozolomide
    * Radiographic progression: Patients with GBM/AA must have radiographic progression based on RANO criteria
    * Therapeutic surgical resection of GBM/AA required as part of routine clinical care
    * Performance status: ECOG 0 or 1
  * Non-Small Cell Lung Cancer (NSCLC) cohort:

    * Previous treatments: No limitations
    * Radiographic progression: Patients must have radiographic progression based on RECIST 1.1 criteria.
    * Measurable Disease
    * Performance Status: ECOG 0 or 1
* Registration - Inclusion Criteria Common to Dose Escalation and Dose Expansion Cohorts:

  * Age >= 18 years old
  * Ability to understand and the willingness to sign a written informed consent document
  * Hemoglobin >= 9.0 g/dL (obtained =< 14 days prior to registration)
  * Leukocytes >= 3.0 x 10^9/L (obtained =< 14 days prior to registration)
  * Absolute neutrophil count >= 1.5 x 10^9/L (obtained =< 14 days prior to registration)
  * Platelets >= 100 x 10^9/L (obtained =< 14 days prior to registration)
  * International normalized ratio (INR) =< 1.5 x upper limit of normal (ULN) (obtained =< 14 days prior to registration)

    * Patients on a stable dose of anti-coagulation therapy will be allowed to participate if they have no signs of bleeding or clotting and the INR/prothrombin time (PT) and partial thromboplastin time (PTT)/activated (a)PTT results are compatible with an acceptable risk-benefit ratio as per the investigator's discretion
  * aPTT =< 1.5 x ULN (obtained =< 14 days prior to registration)

    * Patients on a stable dose of anti-coagulation therapy will be allowed to participate if they have no signs of bleeding or clotting and the INR/PT and PTT/aPTT results are compatible with an acceptable risk-benefit ratio as per the investigator's discretion
  * Total bilirubin =< 1.5 x ULN and =< 3 mg/dL for patients with Gilbert's disease (obtained =< 14 days prior to registration)
  * Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN or =< 5 x ULN if due to liver involvement by tumor (obtained =< 14 days prior to registration)
  * Creatinine =< 1.5 x ULN or estimated glomerular filtration rate (estimated glomerular filtration rate [eGFR]) >= 60 mL/minute (obtained =< 14 days prior to registration)
  * Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only
  * Provision of signed and dated written informed consent prior to any study specific procedures, sampling, and analyses
  * Willingness to provide mandatory blood specimens for correlative research
  * Willingness to return to enrolling institution for follow-up (during the active monitoring phase of the study i.e., active treatment and clinical follow-up)
  * Male and female patients of child bearing potential must be willing to use contraception, (i.e., condoms, birth control) while on study and until 3 months after the last dose of study drug is taken
  * Must be willing to take light-protective measures during the study and for 2 weeks after their last dose of WSD0922-FU
  * Must have a minimum life expectancy of >= 3 months
  * Must be stable on no more than 2 mg of dexamethasone (or equivalent steroids) per day. Steroid dose adjustments should be minimized during cycle 1 of therapy. Patients enrolling to the BTP expansion cohort do not have any restrictions on current steroid/dexamethasone dosing.
  * Must not take enzyme-inducing anticonvulsants treatment for at least 2 weeks prior to enrollment. Patients on enzyme-inducing anticonvulsants will be changed to non-enzyme inducing anticonvulsants
  * Strong inducers and strong inhibitors of CYP3A should be discontinued at least 14 days prior to registration
  * Willingness to provide mandatory tissue specimens for correlative research (BTP cohort only)

Exclusion Criteria:

* Registration - Exclusion Criteria for Dose Escalation and Dose Expansion

  * Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

    * Pregnant persons
    * Nursing persons
    * Persons of childbearing potential who are unwilling to employ adequate contraception
  * Any of the following prior therapies:

    * Any cytotoxic chemotherapy or other anticancer drugs for the treatment of advanced NSCLC from a previous treatment regimen =< 14 days prior to registration
    * In patients with NSCLC, treatment with an EGFR TKI (e.g., erlotinib, gefitinib, afatinib or osimertinib) must be discontinued prior to registration. Additionally, prior EGFR TKI therapy must be discontinued within 8 days or 5 half-lives, whichever is longer, prior to study therapy initiation. If sufficient wash-out time has not occurred due to schedule or PK properties, an alternative appropriate wash-out time based on known duration and time to reversibility of drug related adverse events could be agreed upon by the Investigator and Wayshine)
    * Radiation therapy to the brain =< 12 weeks prior to registration
    * Patients with GBM/AA must not have received (i) nitrosoureas within 42 days of registration, (ii) any chemotherapy or experimental therapy within 28 days or 5 half-lives, whichever is longer, prior to registration
    * Patients with GBM/AA must not have received prior anti-EGFR or EGFRvIII therapies (erlotinib, gefitinib, afatinib, osimertinib, ABT-414, ABBV-221, AMG-595, AMG-596 etc.)
    * Patients with GBM/AA who have been treated with bevacizumab within the last four months are not eligible
    * Received prior systemic biologic therapy (CAR-T, anti-PD-1 / anti-PD-L1, anti-CTLA-4, etc.) within 28 days prior to registration.
  * Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol. Screening for chronic conditions is not required
  * Subjects who are human immunodeficiency virus (HIV), hepatitis virus B (HBV), and/or hepatitis virus C (HCV) positive
  * Uncontrolled inter-current illness including, but not limited to:

    * Symptomatic CNS complications that require urgent neurosurgical or medical (e.g. mannitol) intervention
    * Seizures requiring a change in anti-epileptic medications (addition of new anti-epileptic or increase in dose) =< 2 weeks of registration
    * Known intracranial hemorrhage which is unrelated to tumor
    * Significant medical or psychiatric illness that would interfere with compliance and ability to tolerate treatment as outlined in the protocol
    * Illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers and carcinoma-in-situ of the cervix. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for more than three years prior to registration
* Any of the following cardiac criteria:

  * A marked baseline prolongation of QT/corrected QT (QTc) interval
  * (e.g., repeated demonstration of a QTc interval > 480 milliseconds (ms) (Common Terminology Criteria for Adverse Events [CTCAE] grade 1) using Fridericia's QT correction formula
  * A history of additional risk factors for torsade de pointes (TdP) (e.g., heart failure, hypokalemia, family history of long QT syndrome)
  * The use of concomitant medications that prolong the QT/QTc interval
* Patients confirmed to have a cis double mutation (Del19/T790M or L858R/T790M) or cis triple mutation (Del19/T790m/C797S or L858R/T790M/C797S)
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease. History of hypersensitivity to active or inactive excipients of WSD0922-FU or drugs with a similar chemical structure or class to WSD0922-FU
* Refractory nausea and vomiting if not controlled by supportive therapy, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of WSD0922-FU
* Inadequate bone marrow reserve or organ function
* Patients with NSCLC LM who are unable to undergo collection of CSF
* Patients who are unable to tolerate dairy (GBM/AA cohort only). This is to ensure that patients on this cohort can participate in the food effect study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2031-02-06 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose | Up to 28 days
  The RP2D is either the maximum tolerated dose (MTD) or the highest dose tested (in the case that none of the doses are deemed higher than the MTD), whichever is higher.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 4-6 weeks after study completion
  Assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Overall response rate | Up to 5 years
  The overall response rate will be defined as the number of patients with a partial response (PR) or complete response (CR) that is confirmed in consecutive evaluations (at least 8 weeks apart) divided by the total number of evaluable patients. A 95% confidence interval will also be constructed using the properties of the binomial distribution.
Duration of response (DOR) | From the first occurrence of a PR (or better) and progression, assessed up to 5 years
  Duration of response is defined as the number of days between a patient's first occurrence of a PR (or better) and progression. If a patient goes off study prior to progression (for another reason) then they will be censored at that time. A time to event analysis will be performed utilizing the Kaplan-Meier method which will yield a median DOR.
Progression Free Survival (PFS) | From study entry to disease progression, assessed up to 5 years
  A patient's progression free survival time is the number of days between study entry and disease progression. These data will be analyzed utilizing the Kaplan-Meier method which will yield a median PFS time.

OTHER OUTCOMES:
Pharmacokinetic (PK) analysis (Dose escalation cohort) - AUCs | Day 1 Cycle 1 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual area under curves (AUCs) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics, AUC will then be tested for association changes in responses.
Pharmacokinetic (PK) analysis (Dose escalation cohort) - AUCs | D15 Cycle 1 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual area under curves (AUCs) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics, AUC will then be tested for association changes in responses.
Pharmacokinetic (PK) analysis (Dose escalation cohort) - AUCs | D1 Cycle 2 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual area under curves (AUCs) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics, AUC will then be tested for association changes in responses.
Pharmacokinetic (PK) analysis (Dose escalation cohort) - AUCs | Pre-dose at end of study (EOS) - each cycle is 28 days
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual area under curves (AUCs) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics, AUC will then be tested for association changes in responses.
Pharmacokinetic (PK) analysis (Dose escalation cohort) - Clearance (CL) | Day 1 Cycle 1 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual clearance (CL) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics,as well as the observed Cmax, will then be tested for association changes in responses.
Pharmacokinetic (PK) analysis (Dose escalation cohort) - Clearance (CL) | D15 Cycle 1 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual clearance (CL) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics,as well as the observed Cmax, will then be tested for association changes in responses.
Pharmacokinetic (PK) analysis (Dose escalation cohort) - Clearance (CL) | D1 Cycle 2 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual clearance (CL) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics,as well as the observed Cmax, will then be tested for association changes in responses.
Pharmacokinetic (PK) analysis (Dose escalation cohort) - Clearance (CL) | Pre-dose at end of study (EOS) - each cycle is 28 days
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual clearance (CL) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics,as well as the observed Cmax, will then be tested for association changes in responses.
PK analysis (Cohort I) - AUC | D1 of cycles 1 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual area under curves (AUCs) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics, AUC will then be tested for association changes in responses.
PK analysis (Cohort I) - AUC | D1 of cycle 2 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual area under curves (AUCs) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics, AUC will then be tested for association changes in responses.
PK analysis (Cohort I) - Clearance (CL) | Pre-dose D1 of cycles 3 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual clearance (CL) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics,as well as the observed Cmax, will then be tested for association changes in responses.
PK analysis (Cohort I) - Clearance (CL) | Pre-dose D1 of cycles 4 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual clearance (CL) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics,as well as the observed Cmax, will then be tested for association changes in responses.
PK analysis (Cohort II) - AUC | Day 1 of cycle 0
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual area under curves (AUCs) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics, AUC will then be tested for association changes in responses.
PK analysis (Cohort II) - AUC | Pre-dose D1 of cycles 3 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual area under curves (AUCs) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics, AUC will then be tested for association changes in responses.
PK analysis (Cohort II) - AUC | Pre-dose D1 of cycles 4 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual area under curves (AUCs) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics, AUC will then be tested for association changes in responses.
PK analysis (Cohort II) - Clearance (CL) | Day 1 of cycles 1 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual clearance (CL) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics,as well as the observed Cmax, will then be tested for association changes in responses.
PK analysis (Cohort II) - Clearance (CL) | Day 1 of cycles 2 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual clearance (CL) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics,as well as the observed Cmax, will then be tested for association changes in responses.
PK analysis (Cohort II) - Clearance (CL) | Pre-dose day 1 of cycles 3 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual clearance (CL) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics,as well as the observed Cmax, will then be tested for association changes in responses.
PK analysis (Cohort II) - Clearance (CL) | Pre-dose day 1 of cycles 4 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual clearance (CL) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics,as well as the observed Cmax, will then be tested for association changes in responses.
PK analysis (Cohort III) - AUC | Days 1 and 4 of cycles 0
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual area under curves (AUCs) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics, AUC will then be tested for association changes in responses.
PK analysis (Cohort III) - AUC | Day 1 of cycle 2 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual area under curves (AUCs) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics, AUC will then be tested for association changes in responses.
PK analysis (Cohort III) - AUC | Pre-dose day 1 of cycles 3 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual area under curves (AUCs) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics, AUC will then be tested for association changes in responses.
PK analysis (Cohort III) - AUC | Pre-dose day 1 of cycles 4 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual area under curves (AUCs) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics, AUC will then be tested for association changes in responses.
PK analysis (Cohort III) - Clearance (CL) | Days 1 and 4 of cycles 0
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual clearance (CL) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics,as well as the observed Cmax, will then be tested for association changes in responses.
PK analysis (Cohort III) - Clearance (CL) | D1 of cycle 2 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual clearance (CL) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics,as well as the observed Cmax, will then be tested for association changes in responses.
PK analysis (Cohort III) - Clearance (CL) | Pre-dose day 1 of cycles 3 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual clearance (CL) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics,as well as the observed Cmax, will then be tested for association changes in responses.
PK analysis (Cohort III) - Clearance (CL) | Pre-dose day 1 of cycles 4 (each cycle is 28 days)
  A population pharmacokinetic model will be developed utilizing the pharmacokinetic time points collected, and then used to estimate individual clearance (CL) of WSD0922. The pharmacokinetic will be evaluated by the model, along with other participant factors that may explain the inter-participant variability in pharmacokinetics,as well as the observed Cmax, will then be tested for association changes in responses.
Proteomic analysis | Up to 5 years
  Partial least squares regression will be used to perform unbiased correlations of network-level signaling data acquired from patient samples with patient phenotypic data or to drug distribution data.

CONTACTS AND LOCATIONS:
Overall Officials: Sani H. Kizilbash, M.D., M.P.H., Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials